CLINICAL TRIAL: NCT00005988
Title: A Phase I Open-Label, Safety Study of Haploidentical Bone Marrow Transplantation (BMT) After Ex Vivo Treatment of Bone Marrow With Anti-B7.1 and Anti-B7.2 Antibodies
Brief Title: Bone Marrow Transplantation With Specially Treated Bone Marrow in Treating Patients With Hematologic Cancer That Have Not Responded to Previous Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eva C. Guinan, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-205; P30CA006516 (NIH); GENE-C9909-38; NCI-G00-1801; CDR0000067977 (Other: other)
Record Dates: First submitted 2000-07-05; First posted 2004-05-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myeloma
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; chronic myelomonocytic leukemia; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; refractory cytopenia with multilineage dysplasia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neoplasms, Plasma Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Multiple Myeloma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Leukemia, Myelomonocytic, Chronic; Dendritic Cell Sarcoma, Interdigitating | interventions — Cyclophosphamide; Cyclosporine; Leucovorin; Methotrexate; Methylprednisolone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- in vitro-treated bone marrow transplantation (Experimental): * Donor bone marrow will be harvested on Day -2
  * Bone Marrow incubated with irradiated recipient cells and anti-B7.1 and anti-B7.2 for 36 hours.
  * Bone marrow will be infused intravenously
  * Cyclophosphamide will be administered IV once daily
  * Total Body Irradiation (TBI) will be delivered per institutional practice
  * Methylprednisolone will be administered IV as 4 doses separated by 12 hours,
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: leucovorin calcium; Drug: methotrexate; Drug: methylprednisolone; Procedure: in vitro-treated bone marrow transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cyclosporine
Drug: leucovorin calcium
Drug: methotrexate
Drug: methylprednisolone
Procedure: in vitro-treated bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Treatment of the donor bone marrow with the patient's white blood cells and a monoclonal antibody may prevent this from happening.

PURPOSE: Phase I trial to study the effectiveness of bone marrow transplantation with specially treated bone marrow in treating patients who have hematologic cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if patients with refractory, high risk hematologic malignancies or bone marrow failure who receive HLA haploidentical bone marrow treated with anti-B7 antibody have normal engraftment. II. Determine if these patients are free of hyperacute graft versus host disease (GVHD), defined as grade D GVHD in the first 10 posttransplant days, when treated with this regimen. III. Determine if these patients have an acceptable incidence of life threatening grade D GHVD in the first 50 posttransplant days following this treatment regimen. IV. Determine the safety and tolerability of this treatment regimen in this patient population.

OUTLINE: This is a multicenter study. Patients undergo leukapheresis to collect white blood cells which are incubated with donor bone marrow cells in the presence of anti-B7.1 and anti-B7.2 antibodies for 36 hours. Patients receive total body irradiation twice daily on days -6 to -3, cyclophosphamide IV daily on days -2 and -1, and methylprednisolone IV every 12 hours for a total of 4 doses on days -2 to 0. Patients are infused with the treated donor bone marrow on day 0. Patients then receive methotrexate IV on days 1, 3, 6, and 11 and leucovorin calcium IV 24 hours after each dose of methotrexate every 6 hours for 3-8 doses each time. Patients also receive cyclosporine IV or orally twice daily on days -2 to 100. Patients are followed every 2 months for 1 year.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤40 years.
* Diagnoses-patients with the following hematologic malignancies and bone marrow failure syndromes:

  * Acute myelogenous leukemia-induction failure, relapse, second or greater complete remission (CR)
  * Acute lymphocytic leukemia-induction failure, relapse, second or greater CR, first CR with t(9;22), t(8;14), or t(4;11)
  * Non-Hodgkin's lymphoma (intermediate or high grade) which has failed to achieve CR with at least two induction regimens, relapse, second or greater CR
  * Multiple myeloma with poor prognostic features (elevated 0-2 microglobulin or high labeling index)
  * Hodgkin's disease in relapse or which fails to achieve CR after two chemotherapy regimens
  * Congenital or acquired bone marrow failure - poorly responsive to or intolerant of current therapy
  * Myelodysplastic syndrome of all subtypes except refractory anemia (RA)
* Patient has a haploidentical family member that meets medical criteria for donation.
* Eligibility for other transplant types:

  * Patient considered likely to have clinical deterioration and rapid disease progression during an unrelated donor search, or
  * Patient who has already had an unproductive donor search or
  * Patient ineligible for or has refused autologous transplant
* Adequate renal and hepatic function for age:

  * Serum creatinine <2 x ULN
  * Alanine aminotransferase (ALT, SGPT) x ULN
  * Aspartate aminotransferase (AST, SGOT) x ULN
  * Total bilirubin 5_2 x ULN except if bilirubin is elevated due to Gilbert's syndrome or hemolytic anemia
* Adequate cardiac and pulmonary function for age.
* ECOG Performance Status 0, 1, or 2 or Lansky performance scale >50% for patients <16 years of age.
* Voluntary witnessed written informed consent. Children will be asked for assent where appropriate.
* The patient, if female, must be post-menopausal, premenarcheal, or sterile, or if the patient is of childbearing potential, she must be practicing a method of birth control considered effective and medically acceptable by the investigator for a minimum of 1 month prior to study entry and at least 2 months after the study end.
* Patient must have undergone successful leukapheresis to obtain adequate antigen presenting cells.
* Any patient who enters the study in a relapse state, with evidence of end organ (pulmonary, renal, or hepatic) toxicity, or with recent recovery from infection, who may potentially have little benefit from this protocol, must have his/her eligibility status discussed with the Principal Investigator.
* Patient must have life expectancy of at least 12 weeks.

Exclusion Criteria

* Eligibility for other transplant types:

  * Patient has family donor who is matched or single antigen mismatched at HLA-A, HLA-B, HLA-DR, and HLA-DQ. Donorrecipient matching must be evaluated via both phenotype and genotype.
  * Patient has available unrelated donor who is matched at HLA-A, HLA-B, and HLA-DR. Donor-recipient matching must be evaluated via both phenotype and genotype.
* Active uncontrolled infection (continued positive blood or soft tissue cultures despite appropriate antibiotic treatment)
* Positive 13-HCG in a female of childbearing potential
* Evidence of HIV infection or known HIV positive serology
* Any prior bone marrow transplant
* A peripheral blood differential count at the time of leukapheresis with greater than 25% blasts. This exclusion criterion is valid only for the first four patients enrolled.
* Patients with Fanconi's anemia

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2001-06-16 (Actual); Study Completion 2002-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of primary graft failure | up to 30 days post-transplant

SECONDARY OUTCOMES:
Incidence of hyperacute GVHD | up to 100 days post-transplant
Incidence of Grade D acute GVHD | up to 50 days post-transplant
Incidence of adverse events | up to 100 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Eva Guinan, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies JK, Gribben JG, Brennan LL, Yuk D, Nadler LM, Guinan EC. Outcome of alloanergized haploidentical bone marrow transplantation after ex vivo costimulatory blockade: results of 2 phase 1 studies. Blood. 2008 Sep 15;112(6):2232-41. doi: 10.1182/blood-2008-03-143636. Epub 2008 Jul 10. PMID 18617635